CLINICAL TRIAL: NCT05389969
Title: Efficiency Of Different Intraoral Scanning Techniques In Orthodontic Patients Before And After Brackets Positioning: A Cross Sectional Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Karam Salim, Master's degree student Cairo university, Cairo University
Other Study IDs: 14422020488903
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Digital Orthodontics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: digital arch scanning — Scanning of the maxillary and mandibular dental arch will be performed for the same group of patients twice. The first time is before bracket positioning using two different scanners and the three different techniques. The second time is after brackets positioning using the same two different scanners and the same three different scanning techniques.
  Then these scans will be compared to by superimposition techniques and linear measurement techniques.

SUMMARY:
A Cross-sectional study, in which we compare the efficiency of different scanning techniques in orthodontic patients before and after brackets positioning.

Scanning of the maxillary and mandibular dental arch will be performed for the same group of patients twice. The first time is before bracket positioning using two different scanners and the three different techniques. The second time is after brackets positioning using the same two different scanners and the same three different scanning techniques.

Then these scans will be compared to by superimposition techniques and linear measurement techniques.

DETAILED DESCRIPTION:
In this study two scanners will be utilized Medit i500 and Trios 3. For each scanner three techniques will be used at two different interventions. One before brackets positioning and the other after bracket positioning. American orthodontics ROTH prescription, 0.022 slot metal brackets will be positioned using direct bonding technique.

Three different scanning techniques will be used: buccopalatal technique, S-shaped technique and palatobuccal technique. The buccopalatal technique (A) involves scanning the arch top side starting from the left second molar then run longitudinally to the contra-lateral one. Then go to the buccal side scan from this right side to the contra-lateral side and then palatal scan. Palatal scan done in two steps first was with counterclockwise movement along the palatal vault and then longitudinal movement in postro-anterior direction.

The S-shaped technique (B) involves scanning the arch starting from the palatal side of the left second molar then moving the scanner tip in alternating palatobuccal and buccopalatal S-shaped movement along the arch to the contra-lateral side. Then scanning the mid area of the palate by longitudinal movement in postro-anterior direction.

The palatobuccal technique (c) done by scanning the arch top side first starting from the left second molar runs longitudinally to the contralateral side. Then start palatal scanning by moving the scanner tip with circular movement in a clockwise direction across the palatal vault from the right-side second molar then along the palate to the contralateral second molar. Then the same circular scanning but in the counterclockwise direction to record the remaining part of the palate staring from the left second molar to the contralateral one. The buccal scan will follow starting from the right second molar then run longitudinally to the contralateral side.

ELIGIBILITY:
Inclusion Criteria:

Adolescent patients.

Fully erupted permanent dentition from second molar to the contra lateral second molar in both jaws.

Exclusion Criteria:

Severe degree of malocclusion that prevent full arch bracket positioning

Dento-facial deformity such as cleft lip/ palate or cranio-facial syndrome.

Severe Skeletal discrepancy in any of the three planes of space.

TMD problem

Limited mouth opening

Presence of crowns or bridges.

Ages: 15 Years to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescent patients with Fully erupted permanent dentition from second molar to the contra lateral second molar in both jaws.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Comparison of repeatability between in-vivo and ex-vivo scans | 2 to 3 weeks

SECONDARY OUTCOMES:
The effect of the type of the scanner on the scanning quality. | 2 to 3 weeks
The effect of the bracket presence on the scanning quality. | 2 to 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided